CLINICAL TRIAL: NCT03602534
Title: Thyroid Dysfunction in Female Patients With Acne Vulgaris: [ Relation to Other Variables ]
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diana Gamal Esmat Fouad Botros, Principle Investigator, Assiut University
Other Study IDs: TDFAV
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Acne Vulgaris; Thyroid Dysfunction
Keywords: acne vulgaris; thyroid dysfunction
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples (serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases with variable acne severity scores: * group will include 50 females
  * Clinical examination including acne grade assessment using Global Acne Grading Scale (GAGS)
  * Assessment of body mass index (BMI)
  * blood serum samples will be collected from all patients to do thyroid function test
- healthy controls: * group will include 29 females
  * Assessment of body mass index (BMI)
  * blood serum samples will be collected from all healthy controls to do thyroid function test

SUMMARY:
Acne is a chronic inflammatory disease of the pilo-sebaceous unit with a multi-factorial etiology. It is one of the most frequent cutaneous diseases, affecting more than eighty percent of the population at some point in their lives .

Endocrine factors especially androgens and steroids are one of multiple factors provoked to be involved in pathogenesis of acne . Thyroid hormones have steroid like action that have many regulatory functions in many body organ functions including skin and pilosebaceous unit. Furthermore, subtle thyroid dysfunction was shown to have a role in many disease conditions.

Thyroid hormone action on sebaceous glands is unclear. In hypothyroid states, sebocytes exhibit reduced rates of secretion that increases with thyroxine administration .

DETAILED DESCRIPTION:
Most of studies about thyroid dysfunction in acne patients focused on adult acne population especially females and searched for presence or absence of associating anti-thyroid antibodies with controversial results .

Some other studies were concerned with the impact of acne treatments as tetracycline, isotretinoin or radiotherapy on thyroid pathologies and dysfunction .

Global Acne Severity Scale (GAGS) is a simple, accurate, fast method for the determination of severity of acne, and it requires no special equipment and is relatively cost-effective. Its personal and interpersonal differences is low and it was first used by Doshi and his colleagues in 1997 in USA .

To the best of knowledge, little is published about thyroid dysfunction in acne female patients of different age categories and correlating thyroid function with other important patient and acne variables as body mass index (BMI) , age (starting from 16 years) , acne type, severity and duration.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acne vulgaris from females only with different ages (starting from 16 years) , BMI groups.

Exclusion Criteria:

* Female patients with clinically diagnosed thyroid disease.
* Female patients receiving isotretinoin or minocycline in the last 6 months
* Female patients who were subject to radiotherapy or surgery in neck region.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * multi centers in Assiut city
  * females only
  * age starts from 16 years
Sampling Method: Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
thyroid hormone level in female acne vulgaris patients | 1 hour
  Peripheral blood samples will be taken , for measurement of thyroid hormone by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Emad Taha, Study Director — Assiut University
Locations (1):
- DGamal, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhate K, Williams HC. Epidemiology of acne vulgaris. Br J Dermatol. 2013 Mar;168(3):474-85. doi: 10.1111/bjd.12149. PMID 23210645
- [Background] Zouboulis CC. [Acne vulgaris. The role of hormones]. Hautarzt. 2010 Feb;61(2):107-8, 110-4. doi: 10.1007/s00105-009-1830-1. German. PMID 20107754
- [Background] Contreras-Jurado C, Lorz C, Garcia-Serrano L, Paramio JM, Aranda A. Thyroid hormone signaling controls hair follicle stem cell function. Mol Biol Cell. 2015 Apr 1;26(7):1263-72. doi: 10.1091/mbc.E14-07-1251. Epub 2015 Feb 5. PMID 25657324
- [Background] Shuster S, Thody AJ. The control and measurement of sebum secretion. J Invest Dermatol. 1974 Mar;62(3):172-90. doi: 10.1111/1523-1747.ep12676782. No abstract available. PMID 4361984
- [Background] Vergou T, Mantzou E, Tseke P, Moustou AE, Katsambas A, Alevizaki M, Antoniou C. Association of thyroid autoimmunity with acne in adult women. J Eur Acad Dermatol Venereol. 2012 Apr;26(4):413-6. doi: 10.1111/j.1468-3083.2011.04084.x. Epub 2011 Apr 27. PMID 21521376
- [Background] Ekiz O, Balta I, Unlu E, Bulbul Sen B, Rifaioglu EN, Dogramaci AC. Assessment of thyroid function and lipid profile in patients with postadolescent acne in a Mediterranean population from Turkey. Int J Dermatol. 2015 Dec;54(12):1376-81. doi: 10.1111/ijd.12547. Epub 2015 Mar 13. PMID 25771990
- [Background] Thomson DB, Grammes CF, Starkey RH, Monsaert RP, Sunderlin FS. Thyroid abnormalities in patients previously treated with irradiation for acne vulgaris. South Med J. 1984 Jan;77(1):21-3. doi: 10.1097/00007611-198401000-00007. PMID 6229881
- [Background] Benjamin RW, Calikoglu AS. Hyperthyroidism and lupus-like syndrome in an adolescent treated with minocycline for acne vulgaris. Pediatr Dermatol. 2007 May-Jun;24(3):246-9. doi: 10.1111/j.1525-1470.2007.00395.x. PMID 17542873
- [Background] Uyar B, Solak A, Saklamaz A, Akyildiz M, Genc B, Gokduman A. Effects of isotretinoin on the thyroid gland and thyroid function tests in acne patients: A preliminary study. Indian J Dermatol Venereol Leprol. 2016 Sep-Oct;82(5):587-8. doi: 10.4103/0378-6323.182794. PMID 27212279
- [Background] Doshi A, Zaheer A, Stiller MJ. A comparison of current acne grading systems and proposal of a novel system. Int J Dermatol. 1997 Jun;36(6):416-8. doi: 10.1046/j.1365-4362.1997.00099.x. No abstract available. PMID 9248884
- [Background] Stewart TJ, Bazergy C. Thyroid autoimmunity in female post-adolescent acne: A case-control study. Dermatoendocrinol. 2017 Dec 12;9(1):e1405198. doi: 10.1080/19381980.2017.1405198. eCollection 2017. No abstract available. PMID 29484104